CLINICAL TRIAL: NCT06860958
Title: Roflumilast as an Adjunct to Antidepressants in Major Depressive Disorder Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98421
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine; Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 30 patients will receive fluoxetine 20 mg/day plus placebo
  Interventions: Drug: Fluoxetine; Drug: Placebo
- Comparative group (Active Comparator): 35 patients will receive fluoxetine 20 mg/day plus roflumilast
  Interventions: Drug: Fluoxetine; Drug: Roflumilast

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine is an antidepressant and belongs to a group of medicines known as selective serotonin reuptake inhibitors (SSRIs)
Drug: Roflumilast — Roflumilast is the first drug targeting PDE4 that was marketed for treatment of chronic obstructive pulmonary disease (COPD) with relatively weak potency inducing nausea and vomiting
  Arms: Comparative group
Drug: Placebo — Placebo
  Arms: Control group

SUMMARY:
Major depressive disorder (MDD) is one of the most common psychiatric disorders with serious socioeconomic consequences on daily life and health care costs. Despite the advent of newer antidepressants that target monoamine pathways, nearly 50% of patients have no response to first-line antidepressant therapy. Thus, a combination of medications with different strategies at the beginning of treatment could provide further therapeutic benefits to MDD patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age greater than 18 years old.
2. Patients with Ham-D score at least 18 with item 1 depressed mood scored 2 or greater are eligible.

Exclusion Criteria:

1. Patients with bipolar I or bipolar II disorder; eating disorders, personality disorders, and mental retardation, current diagnosis anxiety disorders (except for specific phobia), mental disorder due to general medical condition; met criteria for substance dependence or abuse in the previous three months; have a concurrent medical illness or history of seizures that would contraindicate use of the study medication and are receiving Electroconvulsive therapy (ECT).
2. Pregnant women or women not using medically accepted means of birth control are excluded.
3. Persons who score greater than 2 on the suicide item of the Ham-D, or who are judged to have significant suicidal ideation or potential in the view of an investigator, are excluded.
4. Patients who are required to be free of all psychotropic except for escitalopram and anti-inflammatory medications for at least four weeks before study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
The principal measure of the outcome will be the 17-item Ham-D | 2 months
  2. Patients will be assessed by a psychiatrist at baseline, 4, and 8 weeks after starting the medication. The principal measure of the outcome will be the 17-item Ham-D.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt